CLINICAL TRIAL: NCT01258972
Title: TRYTON PIVOTAL IDE Coronary Bifurcation Extended Access Study
Brief Title: Prospective, Single Blind, Rand Controlled Study to Evaluate the Safety & Effectness of Tryton Side Branch Stent Used With DES Treatmt of de Novo Bifurcation Lesions in MB & SB in Native Coronaries
Acronym: TRYTON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tryton Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P-0020
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Atherosclerosis of Native Coronary Artery; Bifurcation Lesions: de Novo Lesions of the Main and Side Branch of Native Coronary Artery
Keywords: Bifurcation lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angioplasty POBA (Active Comparator): Side Branch balloon angioplasty with main branch DES
  Interventions: Device: POBA
- Tryton Side Branch Stent (Experimental): Side Branch treated with Tryton Side Branch Stent with main branch DES
  Interventions: Device: Tryton Side Branch Stent with main branch DES

INTERVENTIONS:
Device: Tryton Side Branch Stent with main branch DES — Tryton Side Branch Stent
  Arms: Tryton Side Branch Stent
Device: POBA — Balloon angioplasty
  Arms: Angioplasty POBA

SUMMARY:
The Tryton Side Branch Stent System has been designed to address the procedural difficulty surrounding treatment of bifurcation lesions and to ensure patency of the side branch with similar performance capabilities (e.g., tracking, radiopacity, coverage and radial strength) that are currently available with conventional coronary stents designed for straight (non bifurcation) lesions.

The Tryton Side Branch Stent is intended to treat and maintain patency in the side branch/carina by providing better ostial side branch conformability and is intended for use in conjunction with currently approved balloon-expandable drug-eluding stents for treatment of the main branch.

DETAILED DESCRIPTION:
The use of drug-eluding stents in the treatment of bifurcation lesions suggests that DES reduces the rate of restenosis int he main branch (5-10%); however, results int he side branch are not optimal. A study of T stenting in true bifurcation lesions showed a restenosis rate int he main branch of approximately 6% using the CYPHER stent. However, the same study demonstrated that the restenosis rate remained high int he side branch (20%) despite stent implantation and when restenosis occurs, it is generally located at the ostium of the side branch. Further, in half the cases where PTCA alone was the intended strategy for the side branch, a side branch stent had to be placed to address sub-optimal procedural results.

These findings are consistent with previous metal stent studies and suggest the best long-term results are obtained when a side branch stent is not placed. This study and others suggest that the outcomes are related to the way the stents sit within in the vessel; and therefore a stent designed specifically for bifurcation lesions will be needed to reduce restenosis rates and improve long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 and ≤ 90 years of age;
* Symptomatic ischemic heart disease (CCS class 1-4, Braunwald Class IB, IC, IIB, IIC, IIIB, IIIC, and/or have objective evidence of myocardial ischemia);
* Acceptable candidate for CABG;
* Intent to treat the side branch of the target bifurcation based on angiographic evaluation;
* The patient is willing to comply with specified follow-up evaluations;
* The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics Committee (MEC) or Institutional Review Board (IRB).
* Planned use of one of the following approved and commercially available drug-eluting stents for subject's index procedure: CYPHER®, ENDEAVOR® RESOLUTE, PROMUS® or PROMUS® ELEMENT, XIENCE™ V or XIENCE PRIME.

General Exclusion Criteria

* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test;
* Patient has had a known diagnosis of STEMI acute myocardial infarction (AMI) within 72 hours preceding the index procedure or >72 hours preceding the index procedure and CK and CK-MB have not returned to within normal limits at the time of procedure;
* Patients with non-STEMI within 7 days prior to index procedure with continued CK-MB elevation;
* Patients with non-target lesion PCI within 7 days prior to index procedure with continued CK-MB elevation;
* Impaired renal function (serum creatinine >2.5 mg/dL or 221 μmol/l) or on dialysis;
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC <3,000 cells/mm3;
* Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or any other significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Patient has received an organ transplant or is on a waiting list for any organ transplant;
* Patient has other medical illness (e.g., cancer, known malignancy, or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
* Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, prasugrel, stainless steel alloy, cobalt-chromium alloy, rapamycin, everolimus, zotarolimus, paclitaxel, and/or contrast sensitivity that cannot be adequately pre-medicated;
* Patient presents with cardiogenic shock or cardiac arrhythmias that create hemodynamic instability;
* Patient in whom a surgical or other procedure is planned within the next year which would require discontinuation of dual antiplatelet therapy;
* Currently participating in another investigational drug or device study or patient inclusion in another investigational drug or device study where the primary endpoint of the study has not been reached.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-12; Primary Completion 2014-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 9 months

SECONDARY OUTCOMES:
In-segment % diameter stenosis of the Tryton SB compared to side branch balloon angioplasty | 9 months

OTHER OUTCOMES:
Periprocedural MI after PCI, CK-MB elevation with value >3X times the upper range limit within the first 48 hrs after PCI | 48 hours post PCI
  Extended Access Registry is the extension of the Prospective multicenter, randomized, controlled study designed to enroll up to 133 subjects treated with the tryton Side Branch Stent with main branch approved DES for treatment of native coronary artery bifurcation disease in lesions >/= 2.5mm RVD

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, M.D., Principal Investigator — Columbia University
Locations (1):
- Jeffery Moses, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grundeken MJ, Collet C, Ishibashi Y, Genereux P, Muramatsu T, LaSalle L, Kaplan AV, Wykrzykowska JJ, Morel MA, Tijssen JG, de Winter RJ, Onuma Y, Leon MB, Serruys PW. Visual estimation versus different quantitative coronary angiography methods to assess lesion severity in bifurcation lesions. Catheter Cardiovasc Interv. 2018 Jun;91(7):1263-1270. doi: 10.1002/ccd.27243. Epub 2017 Aug 24. PMID 28836339
- [Derived] Muramatsu T, Grundeken MJ, Ishibashi Y, Nakatani S, Girasis C, Campos CM, Morel MA, Jonker H, de Winter RJ, Wykrzykowska JJ, Garcia-Garcia HM, Leon MB, Serruys PW, Onuma Y; TRYTON Pivotal IDE Coronary Bifurcation Trial Investigators. Comparison between two- and three-dimensional quantitative coronary angiography bifurcation analyses for the assessment of bifurcation lesions: A subanalysis of the TRYTON pivotal IDE coronary bifurcation trial. Catheter Cardiovasc Interv. 2015 Sep;86(3):E140-9. doi: 10.1002/ccd.25925. Epub 2015 Apr 24. PMID 25914327
- [Derived] Grundeken MJ, Ishibashi Y, Genereux P, LaSalle L, Iqbal J, Wykrzykowska JJ, Morel MA, Tijssen JG, de Winter RJ, Girasis C, Garcia-Garcia HM, Onuma Y, Leon MB, Serruys PW. Inter-core lab variability in analyzing quantitative coronary angiography for bifurcation lesions: a post-hoc analysis of a randomized trial. JACC Cardiovasc Interv. 2015 Feb;8(2):305-314. doi: 10.1016/j.jcin.2014.12.002. PMID 25700754
- [Derived] Genereux P, Kumsars I, Lesiak M, Kini A, Fontos G, Slagboom T, Ungi I, Metzger DC, Wykrzykowska JJ, Stella PR, Bartorelli AL, Fearon WF, Lefevre T, Feldman RL, LaSalle L, Francese DP, Onuma Y, Grundeken MJ, Garcia-Garcia HM, Laak LL, Cutlip DE, Kaplan AV, Serruys PW, Leon MB. A randomized trial of a dedicated bifurcation stent versus provisional stenting in the treatment of coronary bifurcation lesions. J Am Coll Cardiol. 2015 Feb 17;65(6):533-43. doi: 10.1016/j.jacc.2014.11.031. PMID 25677311
- See also: Sponsor website — http://www.trytonmedical.com